CLINICAL TRIAL: NCT04177433
Title: The Use of Intra-articular Corticosteroid Injection to Treat Osteoarthritis of the Carpometacarpal Joint: A Randomized Control Trial
Brief Title: The Use of Intra-articular Corticosteroid Injection to Treat Osteoarthritis of the Carpometacarpal Joint
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00092745
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis of the Carpometacarpal Joint; Thumb Osteoarthritis
Keywords: Basal thumb arthritis; Carpometacarpal arthritis; Steroid injection; Thumb osteoarthritis
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid Injection (Experimental): Pre-filled opaque syringe containing 40 mg (1cc) of depo-medrol combined with 0.5 cc of 1% lidocaine (or 1cc saline + 0.5 cc 1% lidocaine) will be injected in the symptomatic CMC joint using fluoroscopic imaging to ensure injection into the joint. If both CMC joints are symptomatic, the most symptomatic joint will be injected. If both CMC joints are equally symptomatic, the dominant hand will be injected.
  Interventions: Drug: Depo-Medrol Injectable Product
- Saline (Placebo Comparator): Pre-filled opaque syringe containing 0.5 cc of 1% lidocaine (or 1cc saline + 0.5 cc 1% lidocaine) will be injected in the symptomatic CMC joint using ultrasound imaging to ensure accuracy of injected location. If both CMC joints are symptomatic, the most symptomatic joint will be injected. If both CMC joints are equally symptomatic, the dominant hand will be injected.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Depo-Medrol Injectable Product — Corticosteroid
  Arms: Corticosteroid Injection
Drug: Saline — Placebo
  Arms: Saline

SUMMARY:
This randomized clinical trial (RCT) will evaluate 6-month outcomes following intra-articular injections for arthritis of the thumb carpometacarpal (CMC) joint by comparing corticosteroid plus local anesthetic versus saline (placebo) plus local anesthetic.

DETAILED DESCRIPTION:
Background & Significance:

The burden of chronic diseases such as osteoarthritis (OA) is increasing globally, having a major impact on both health services and society. 1,2 The CMC joint of the thumb is the most commonly affected joint in the upper extremity by OA, and may lead to pain, decreased hand function and poor health-related quality of life. 3-6 The prevalence of CMC OA varies depending on the population being studied and is not yet well defined. Haara et al. 6 reported age-adjusted CMC OA prevalence of 7% in men and 15% in women among adults thirty years of age or older in Finland. The ROTTERDAM study7 showed that 67% of the women and 54.8% of the men had OA in at least one hand joint, with 35.8% occurring at the CMC joint. The Framingham Study reported higher prevalence of symptomatic hand OA in women (26.2%) compared to men (13.4%) aged 70 year or older. Symptomatic participants in this cohort had 10% reduced maximal grip strength, reported more difficulty with activities of daily living such as writing, handling, or fingering small objects (odds ratio = 3.4), and increased difficulty lifting over 10-pound objects (odds ratio = 1.7 and 1.6, respectively).8

Treating CMC OA is challenging, since evidence is contradictory. A study looking at the natural history of hand OA over a 6 year period showed variation in pain and functional changes, with half of the population reporting deterioration of symptoms and the other half reporting improvements of outcomes with different treatments. 9 Clinical changes (pain and function) and radiographic progression of CMC OA were not related in this study. 9 Non-operative management (i.e. splints, medications, physiotherapy) is usually the first choice of treatment for symptomatic CMC OA, followed by surgery if failed non-operative management. 3,10 Current non-operative guidelines for treatment of hand OA are based on a combination of research findings and expertise opinion. 11-13 2007EULAR, 2012 American College of Rheumatology and 2014 NICE guidelines recommendations for the treatment of hand OA include general considerations (i.e. clinical presentation, risk factors and associated diseases), non-pharmacological (i.e. splint, education, exercises, thermal modalities), and pharmacological (i.e. pain medications, oral and topical anti-inflammatories, opioids) approaches. 11-13 2007EULAR and 2014 NICE also recommend intra-articular corticosteroid injections as an adjunct treatment if patients didn't respond to other treatment approaches, even though evidence is weak.11,13

Effectiveness of guided intra-articular injections for CMC OA evidence is inconsistent. There is only one published RCT looking specifically at efficacy of corticosteroid injections in CMC OA that found no clinical benefit from intra-articular corticosteroid injection to moderate to severe CMC OA compared with placebo injection. This study ended earlier due to recruitment issues and is underpowered to detect true differences between groups. 14 A meta-analysis investigating intra-articular injections of corticosteroids or hyaluronic acid in thumb OA stated that corticosteroids may be helpful in decreasing pain and hyaluronic acid in improving pulp pinch force in a period of 5 to 6 months. 15 Due to high heterogeneity of included studies in this meta-analysis, the evidence is still inconclusive. Another RCT compared the efﬁcacy of intra-articular hyaluronic acid and corticoid injections in CMC OA and found that both study groups had decreased pain and improved function when compared to baseline data, with no significant differences between groups. 16 A recent systematic review on non-surgical therapies for hand OA found inconsistent evidence when comparing intra-articular steroids and placebo. 17 They found three RCTs comparing intra-articular steroids to placebo, with two studies showing no difference and one study showing significant improvement in pain with movement between groups.17

Based on the lack of strong evidence regarding the use of guided corticosteroid injections to treat CMC OA, this randomized clinical trial (RCT) will compare 6-months outcomes following fluoroscopic guided injections of corticosteroid plus local anesthetic or saline (placebo) plus local anesthetic in adult participants with carpometacarpal osteoarthritis (OA).

Our hypothesis is that participants undergoing guided intra-articular corticosteroid injections will have better outcomes in the short -term, but not at the long term when compared to the saline group.

Research Design & Methods:

Design: Randomized Control Trial Sample Size: Sample size was calculated based on repeated measures ANOVA model with 2 groups and 4 time points (longitudinal approach), and group effect (between subject effect) were examined for power analysis. Effect size (Cohen's f) was considered from f=0.10 (small effect) to f=0.40 (large effect) increased by 0.05. Few different correlations among repeated measures were considered (r=0.3 to 0.6 by 0.1). Based on effect size f=0.25 (medium effect), approximately 62 to 90 participants will be required as total sample size, with approximately 31to 45 participants per group.

Enrollment Procedures: Eligible participants presenting to primary care, rheumatologists or a surgical consult will be introduced to the study. If the participant expresses interest, the participant will complete the contact information form (assent to contact) and the Research Coordinator will be notified. The Research Coordinator will contact the participant to discuss the study in detail, obtain informed consent and book a baseline assessment.

Baseline Evaluation: Consented participants will undergo a baseline assessment with the research coordinator who will be blinded to the treatment allocation. The assessment will consist of 1) Quick-DASH, 2) Brief Michigan Hand Outcomes Questionnaire (Brief MHQ), 3) grip and pinch strength using a handheld dynamometer, 4) socio-demographics (age, gender, height, weight, handedness, smoking status, work/recreational sports information, duration of symptoms, type of onset (insidious / traumatic) data). The participant will also complete the Visual Analogue Scale (VAS) for pain intensity (rest and movement), and concomitant treatments form (medications, splints, physiotherapy,…).

Randomization:

Participants will be randomized to one of the two groups once eligibility is confirmed and participant is agreeable to be part of the study: Group A (intra-articular corticosteroid injection + local anesthetic) or Group B (saline injection + local anesthetic). The randomization sequence will be computer-generated in uneven blocks. Randomization codes will be stored in opaque sequentially numbered envelopes and will be opened at baseline assessment session. Participants and outcomes assessor will be blinded to the type of injection they will be receiving.

Interventions:

* Fluoroscopic Guided Intra-articular Corticosteroid Injection plus local anesthetic: Pre-filled opaque syringe containing 40 mg (1cc) of depo-medrol combined with 0.5 cc of 1% lidocaine (or 1cc saline + 0.5 cc 1% lidocaine) will be injected in the symptomatic CMC joint using fluoroscopic imaging to ensure injection into the joint. If both CMC joints are symptomatic, the most symptomatic joint will be injected. If both CMC joints are equally symptomatic, the dominant hand will be injected. The surgeon and the participant will be blinded to the injection content.
* Fluoroscopic Guided Intra-articular Saline Injection plus local anesthetic: Pre-filled opaque syringe containing 0.5 cc of 1% lidocaine (or 1cc saline + 0.5 cc 1% lidocaine) will be injected in the symptomatic CMC joint using ultrasound imaging to ensure accuracy of injected location. If both CMC joints are symptomatic, the most symptomatic joint will be injected. If both CMC joints are equally symptomatic, the dominant hand will be injected. The surgeon and the participant will be blinded to the injection content.

Follow-ups:

Follow-up research assessments will occur at:

• 6 weeks, 3- and 6-months: Assessment will be done by the research coordinator and will include 1) Quick-DASH, 2) Brief MHQ, 3) Grip and Pinch strength, 4) Pain at rest and with movement, 5) Concomitant treatments tracking.

The outcome assessor will be blinded to group allocation at all assessments points.

Outcomes/ Outcome Measures:

* Primary:

  o Pain with movement at 3 months- Pain will be assessed using Visual Analogue Scale (VAS) where zero equaled no pain and 10 the worst possible pain.18,19 VAS is a reliable and valid method of measuring patient-reported pain and a minimal difference of 20 mm (20%) among groups will be considered clinically important.20-22
* Secondary Outcomes:

  * Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) Questionnaire: it's a 11-item, patient-reported questionnaire that measures the function and psychosocial impact of upper extremity musculoskeletal conditions in patients' quality of life. It is scored between 0 (no disability) and 100(very disable).23 The Quick-DASH has been widely used in clinical practice and research as a valid, reliable and responsive tool to measure treatment outcomes from the patient's perspective after upper limb injuries.24 The minimal important change expected is a 10-point difference in mean DASH score among groups.24
  * Brief Michigan Hand Outcomes Questionnaire (Brief MHQ): It is a 12-item self-administered questionnaire that assess function, appearance, pain, and satisfaction in patients with hand and wrist conditions and injuries, including arthritis.
  * Pinch Strength: Pinch strength will be measured with a mechanical pinch gauge that is a reliable and valid method to detect difference in thumb strength.26 Pinch strength will be measured using the following standard positions: 1) Tip pinch: pinch between the thumb and index finger, and 2) Tripod pinch: pinch between the thumb, index and middle fingers.26 A minimal difference of 0.33 kg for tip and 0.35 kg for tripod pinch among groups will be considered clinically important.26

Statistical Analysis: Statistical analysis will use Intention-to-Treat approach with all outcomes attributed to the assigned group. Descriptive statistics will be used for group comparisons with independent t-tests for continuous and Pearson Chi-square or Fisher's Exact tests for categorical variable at baseline and for possible complications/adverse events. Linear Mixed Modeling (LMM), adjusted for gender and employment, will compare pain, Quick-Dash, Brief MHQ and pinch strength between groups over the 6-months evaluation period. The level of significance will be set at α=0.05. Statistical analysis will use the following software: SPSS version 25.0, SAS version 9.4, and R version 3.5.2.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years old or older at recruitment
* Present clinical and radiographic signs of thumb CMC OA using the American College of Rheumatology (ACR) criteria for the classification of hand osteoarthritis.

Exclusion Criteria:

* History of inflammatory arthritis
* Previous steroid joint injection to either thumb CMC joint
* Pregnancy or breastfeeding
* Psychiatric illness
* Cognitive impairment, or health conditions that preclude informed consent or receiving the injection
* People who do not speak/read/understand English, have no fixed address or contact, or are unwilling to complete follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain with movement | baseline, 6 weeks, 3 months, 6 months
  Pain will be assessed using Visual Analogue Scale (VAS) where zero equaled no pain and 10 the worst possible pain. a minimal difference of 20 mm (20%) between groups will be considered clinically important.

SECONDARY OUTCOMES:
Change in Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) Questionnaire | baseline, 6 weeks, 3 months, 6 months
  it's a 11-item, patient-reported questionnaire that measures the function and psychosocial impact of upper extremity musculoskeletal conditions in patients' quality of life. It is scored between 0 (no disability) and 100(very disable). The minimal important change expected is a 10-point difference in mean DASH score among groups.
Change in Brief Michigan Hand Outcomes Questionnaire | baseline, 6 weeks, 3 months, 6 months
  Brief Michigan Hand Outcomes Questionnaire (Brief MHQ): It is a 12-item self-administered questionnaire that assess function, appearance, pain, and satisfaction in patients with hand and wrist conditions and injuries, including arthritis.
Change in Pinch Strength | baseline, 6 weeks, 3 months, 6 months
  Pinch strength will be measured with a mechanical pinch gauge that is a reliable and valid method to detect difference in thumb strength. Pinch strength will be measured using the following standard positions: 1) Tip pinch: pinch between the thumb and index finger, and 2) Tripod pinch: pinch between the thumb, index and middle fingers. A minimal difference of 0.33 kg for tip and 0.35 kg for tripod pinch among groups will be considered clinically important.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Hand & Upper Limb Facility, Sturgeon Community Hospital, St. Albert, Alberta, Canada